CLINICAL TRIAL: NCT05994664
Title: The Effects Of Heart Coherence Training On Patients With Vascular Ehlers-Danlos Syndrome (HEARTMATH)
Brief Title: Heart Coherence Training on Vascular Ehlers-Danlos Syndrome Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Southern Star Research (Industry)
Responsible Party: Principal Investigator, Shaine Morris, Associate Professor, Pediatrics-Cardiology, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: H-53424
Record Dates: First submitted 2023-08-09; First posted 2023-08-16 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Vascular Ehlers-Danlos Syndrome
Keywords: Cardiovascular; Mental Health; Heart Rate Variability
MeSH Terms: conditions — Ehlers-Danlos Syndrome, Type IV; Psychological Well-Being | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Trial will have two parallel groups and randomization will be performed at a 1:1 allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group of up to 20 patients will be randomly allocated into an experimental group at a 1:1 ratio intervention to controls. The experimental group will receive all of the preliminary outcome screening with the additional 10-15 minutes of training and advancement on HeartMath techniques as well as continued written and video reinforcement.
  Interventions: Other: Heartmath Intervention
- Control (Placebo Comparator): Group of up to 20 patients will be randomly allocated into a control group at a 1:1 ratio for intervention to controls. The control group will receive all of the preliminary outcome screening and will have weekly virtual sessions that include the 3-step Protocol HRV assessment. After the CG has completed 8 weeks, they will then have access to materials related to the techniques that were taught to the HMI group to allow for therapeutic equality.
  Interventions: Other: Control Group

INTERVENTIONS:
Other: Heartmath Intervention — The participants will all complete baseline surveys and paperwork including signed consent, psychometric surveys, demographic survey, and a brief, open-ended questionnaire about their feelings about living with VEDS. During the initial visit for the intervention group the same assessment will be included, however, they will also receive 10-15 of instruction on a basic Heartmath technique. Group participants will be asked to complete 5-10 minutes of HeartMath techniques 2x daily. Participants from both groups will have weekly virtual sessions that include the 3-step Protocol HRV assessment. However, each week the intervention group will receive an addition 10-15 minutes of training and advancement on HeartMath techniques as well as continued written and video reinforcement.
  Arms: Intervention
Other: Control Group — The participants will all complete baseline surveys and paperwork including signed consent, psychometric surveys, demographic survey, and a brief, open-ended questionnaire about their feelings about living with VEDS. The initial visit will include an HRV assessment using the HeartMath sensor via the 3-step Protocol developed by the HeartMath Institute. Participants from both groups will have weekly virtual sessions that include the 3-step Protocol HRV assessment. After the CG has completed 8 weeks, they will then have access to materials related to the techniques that were taught to the HMI group to allow for therapeutic equality.
  Arms: Control

SUMMARY:
Vascular Ehlers-Danlos Syndrome (VEDS) is caused by pathogenic variants of the COL3A1 gene, resulting abnormal Type III collagen protein. This impacts the body's connective tissue and makes people with VEDS at high risk of spontaneous aortic and arterial rupture, pneumothorax, and hollow organ perforation across the age spectrum. Given this risk and high potential for lethality, VEDS is considered the most severe type of Ehlers-Danlos Syndrome. In addition, many patients experience chronic pain and fatigue, sleep disturbances, and mental health challenges. As is the case for many patients with chronic illness, stress, anxiety, and depression are often present over the course of the disease. Despite the antecedent, stress and anxiety trigger a sympathetic nervous system (SNS) response in the body, which, over a period of time, can have detrimental effects both physiologically and psychologically for patients. Recent studies have begun to use biofeedback techniques to teach patients non-pharmacological strategies for managing their autonomic nervous system. One such program, Heartmath®, has been successful in helping patients lower stress, anxiety, and systolic blood pressure. This pilot trial was established to assess the effectiveness of a virtually based heart coherence program in a population with a chronic aortopathy in an effort to establish a larger, multi-provider program that also encompasses other cardiovascular populations.

DETAILED DESCRIPTION:
Vascular Ehlers Danlos Syndrome (VEDS) is caused by pathogenic variants of the COL3A1 gene, resulting abnormal Type III collagen protein. This impacts the body's connective tissue and makes people with VEDS at high risk of spontaneous aortic and arterial rupture, pneumothorax, and hollow organ perforation across the age spectrum. Given this risk and high potential for lethality, VEDS is considered the most severe type of Ehlers-Danlos Syndrome. In addition, many patients experience chronic pain and fatigue, sleep disturbances, and mental health challenges. As is the case for many patients with chronic illness, stress, anxiety, and depression are often present over the course of the disease. Despite the antecedent, stress and anxiety trigger a sympathetic nervous system (SNS) response in the body, which, over a period of time, can have detrimental effects both physiologically and psychologically for patients. For patients with already compromised cardiovascular systems, the dysregulation of their nervous system can potentially be detrimental to their mental and physiological health, as well as their overall quality of life.

Recent studies have begun to use biofeedback techniques to teach patients non-pharmacological strategies for managing their autonomic nervous system. One such program, Heartmath®, has been successful in helping patients lower stress, anxiety, and systolic blood pressure.

Our primary aim of this study is to evaluate the effects of an 8 week, virtually-based heart coherence training program (HCTP) with the use of wearable, biofeedback technology. The goal is to perform a randomized-controlled pilot study to assess effect estimates on multiple outcomes in an effort to establish a foundation for a larger, longitudinal trial.

The objective is to:

1. Randomize 20 patients with Vascular Ehlers-Danlos Syndrome from ages 12 -45 years to current status and care (controls) versus a biofeedback intervention of additional training and advancement on HeartMath techniques, then
2. Allow the control group subjects to then have access to materials related to the techniques that were taught to the HMI group to allow for therapeutic equality. The investigators will then compare outcomes between both the intervention and control groups, and between the baseline and post-intervention states. Specific outcome measures will include ambulatory blood pressure, heart rate variability, coherence ratio, mean heart rate, quality of life/mental health assessment: health-related quality of life, depression and anxiety screening scales.

Our hypothesis is that individuals with VEDS undergoing a supervised HCTP will demonstrate improvements in ambulatory blood pressure, heart rate variability, and mental health survey measures.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be diagnosed with Vascular Ehlers-Danlos Syndrome verified by a mutation of the COL3A1 gene
* Ages 12-45 year at the time of enrollment
* Access to a smartphone as well as an additional device with camera and microphone
* Stable internet access
* English speaking

Exclusion Criteria:

* Non-English speakers
* Any conditions or developmental delays limiting the ability to utilize technology or follow directions.

Ages: 12 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Mean Overall Systolic Blood Pressure | 3 Months
  Comparing baseline to post-intervention overall systolic blood pressure in percent

SECONDARY OUTCOMES:
Mean systolic blood pressure | 3 Month
  mmHg, range 70-200, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Mean Diastolic blood pressure | 3 Month
  mmHg, range 20-150, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Nocturnal systolic blood pressure | 3 Month
  mmHg, range 70-200, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile, nocturnal reading
Nocturnal Diastolic blood pressure | 3 Month
  mmHg, range 20-150, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile, nocturnal reading
Diurnal Systolic blood pressure | 3 Month
  mmHg, range 70-200, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile, diurnal reading
Diurnal Diastolic blood pressure | 3 Month
  mmHg, range 20-150, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile, diurnal reading
Daily Systolic blood pressure | 3 Month
  mmHg, range 70-200, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Daily Diastolic blood pressure | 3 Month
  mmHg, range 20-150, both low and high are abnormal, goal is age, sex and height-based, goal 10-50 percentile
Coherence Percentage | 3 Months
  Between 0.04-0.24 Hz (3-15 cycles per min), The more stable and regular the heart rhythm frequency is the higher the coherence. Percent ranges from 0.5 Basic good beginner level, 1.0 Good, 2.0 Very Good, 3.0+ Excellent. The higher the percentage the better.
Heart rate variability | 3 Months
  Consists of beat to beat changes in heart rate measured by values below 50 ms are classified as unhealthy, 50-100 ms have compromised health, and above 100 ms are classified as healthy.
Mean Heart Rate | Measured at baseline and follow up visit (at 12 weeks)
  Measured for 24 hrs, range of 60-100 bpm
Nocturnal Heart Rate | Measured at baseline and follow up visit (at 12 weeks)
  Adolescent: 50-90 bpm and Adult: 40-50 bpm, measured for 24 hours
Diurnal Heart Rate | Measured at baseline and follow up visit (at 12 weeks)
  Adolescent: 60-100 bmp and Adult: 60-100 bmp, measured for 24 hours
Quality of Life Scale (QOLS) (ages 19-21 y) | 3 Months
  16 items, each with 7 point Likert, higher is worse
Pediatric Quality of Life Scale (PedsQL) scale scores | 3 Months
  reported in 3 domains, each reported on Likert scale, scaled to 0-100 scale, lower is worse
GAD-7 | 3 Months
  Seven-item questionnaire that detects generalized anxiety disorder and the severity of the anxiety. Total score for the seven items ranges from 0 to 21. The higher the score the worse; cut off score is 8.
PSC | 3 Months
  The Pediatric Symptom Checklist (PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. A positive score on the PSC or Y-PSC suggests the need for further evaluation by a qualified health. PSC-35-Youth, English & Spanish cut off score is, 30 or higher. In a Mexican-American sample, a cutoff score of 12 was shown to be most sensitive.
PSC-Y | 3 Months
  The Pediatric Symptom Checklist (PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. A positive score on the PSC or Y-PSC suggests the need for further evaluation by a qualified health. PSC-35-Youth, English & Spanish cut off score is, 30 or higher. In a Mexican-American sample, a cutoff score of 12 was shown to be most sensitive.PSC Subscales:Attention Problems, Internalizing Problems, Externalizing Problems
PSC-Y Attention Subscale | 3 Months
  The Pediatric Symptom Checklist (PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. A positive score on the PSC or Y-PSC suggests the need for further evaluation by a qualified health. PSC-35-Youth, English & Spanish cut off score is, 30 or higher. In a Mexican-American sample, a cutoff score of 12 was shown to be most sensitive.
  PSC Subscales:Attention Problems Subscale: Children with subscores greater than or equal to 7 usually have significant impairments in attention.
PSC-Y Internalizing Problems Subscale | 3 Months
  The Pediatric Symptom Checklist (PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. A positive score on the PSC or Y-PSC suggests the need for further evaluation by a qualified health. PSC-35-Youth, English & Spanish cut off score is, 30 or higher. In a Mexican-American sample, a cutoff score of 12 was shown to be most sensitive.
  PSC Subscales:
  Internalizing Problems Subscale: Children with subscores greater than or equal to 5 usually have significant impairments with anxiety or depression.
PSC-Y Externalizing Problems Subscale | 3 Months
  The Pediatric Symptom Checklist (PSC) is a 35 item questionnaire that helps identify and assess changes in emotional and behavioral problems in children. A positive score on the PSC or Y-PSC suggests the need for further evaluation by a qualified health. PSC-35-Youth, English & Spanish cut off score is, 30 or higher. In a Mexican-American sample, a cutoff score of 12 was shown to be most sensitive.
  PSC Subscales:
  Externalizing Problems Subscale: Children with subscores greater than or equal to 7 usually have significant problems with conduct.
PROMIS Pediatric Self- Reported Psychological Stress | 3 Months
  PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. On the T-score metric, A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Better health is a lower score and worse health scores higher.
PROMIS Parent Proxy Reported Psychological Stress- Parent Proxy | 3 Months
  PROMIS scores have a mean of 50 and standard deviation (SD) of 10 in a referent population. On the T-score metric, A score of 40 is one SD lower than the mean of the reference population. A score of 60 is one SD higher than the mean of the reference population. Higher score is worse health.
The PROMIS Adult Depression SF v1.0 8a | 3 Months
  Adult measure is the 8-item PROMIS Depression Short Form v1.0 8a questionnaire that assesses the pure domain of depression in individuals age 18 and older.
  A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like depression, a T-score of 60 is one SD worse than average. By comparison, a depression T-score of 40 is one SD better than average.
The PROMIS Pediatric Depression SF V2.0 8a | 3 Months
  The PROMIS Short Form v2.0 - Depression 8a questionnaire includes 8 questions related to depressed mood in the past 7 days for ages 8-17.
  A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like depression, a T-score of 60 is one SD worse than average. By comparison, a depression T-score of 40 is one SD better than average.
The PROMIS Parent Proxy Depression SF v2.0 6a | 3 Months
  The PROMIS Short Form v2.0 - Depression 6a questionnaire includes 6 questions related to depressed mood in the past 7 days for parents serving as proxy reporters for their child (youth ages 5-17).
  A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like depression, a T-score of 60 is one SD worse than average. By comparison, a depression T-score of 40 is one SD better than average.

CONTACTS AND LOCATIONS:
Overall Officials: Shaine A Morris, MD, MPH, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States